CLINICAL TRIAL: NCT06278974
Title: A Comparative Study on the Clinical Efficacy, Quality of Life, and Cost of Use of Peripheral Defocus Spectacles, Frame Glasses, and Orthokeratology Lenses in Myopic Children and Adolescents
Brief Title: Comparing Myopia Treatments in Youth: Defocus Spectacles, Glasses, and Ortho-K
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PDSFGOCLMC-2023-001
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: Myopia; Cost-effectiveness Analysis; Quality of Life
Keywords: Myopia; youth; glasses
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control Group1: This group includes children and adolescents who are correcting myopia using peripheral defocus spectacles. These spectacles are a novel corrective measure, designed to control myopia progression by creating a defocus zone around the periphery of the lenses.
- Control Group2: This group consists of children and adolescents using orthokeratology lenses for myopia correction. Orthokeratology lenses are specially designed rigid contact lenses worn overnight to temporarily reshape the cornea, aiming to reduce dependency on glasses or contact lenses during the day.
- Control Group3: This group includes children and adolescents who are using standard single-vision frame glasses for myopia correction.

SUMMARY:
The research project titled "A Comparative Study on the Clinical Efficacy, Quality of Life, and Cost of Use of Peripheral Defocus Spectacles, Frame Glasses, and Orthokeratology Lenses in Myopic Children and Adolescents" aims to evaluate different non-surgical myopia correction methods in children. It focuses on assessing the impact of peripheral defocus spectacles, frame glasses, and orthokeratology lenses on the quality of life, clinical effectiveness, and costs associated with each method. The study is a prospective cohort study involving 300 children aged 13-17 years with myopia ranging from -1.00D to -6.00D. It aims to compare the psychological, social, and educational aspects of these correction methods, alongside their costs and clinical outcomes over a period of one year.

DETAILED DESCRIPTION:
The research project "Comparison of the clinical effect, quality of life and cost of using defocusing glasses, frame glasses and orthokeratology glasses in children and adolescents with myopia" aims to explore the impact of different myopia correction methods on children and adolescents. Myopia is one of the most common eye diseases in the world, especially in East Asia, where the incidence of myopia is extremely high. With the development of China's economy and the increasing pressure of children's education, the problem of myopia is becoming more and more serious, and parents and teenagers lack sufficient information and evidence for choosing the most suitable correction methods.

This study will compare the defocus frame glasses, ordinary monopteral frame glasses and orthokeratology glasses. The defocusing frame glasses are a new correction method, showing potential in controlling the length of the eye axis. Ordinary single-frame glasses are the most commonly used and economical choice; The orthokeratology lens is a kind of hard contact lens worn at night, which is in fast growing demand in the Chinese market.

The main objectives of the study include:

Quality of life assessment: To explore the impact of different correction methods on adolescents' daily life, learning, movement, appearance, mental health and social activities.

Use cost analysis: Compare the purchase cost, maintenance cost and replacement frequency of defocusing frame glasses, monopter frame glasses and orthokeratology glasses to assess the economic burden of long-term use.

In addition, the study will comprehensively evaluate the differences in clinical effectiveness, quality of life and cost of use of these correction methods, providing parents and adolescents with more comprehensive and objective information to help them make more informed choices.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 13-17 years.
* Myopia between -1.00D and -6.00D; astigmatism <±1.5D; best corrected visual acuity ≥1.0.
* No prior use of peripheral defocus spectacles, single-vision frame glasses, or orthokeratology lenses (meaning first-time wearers).
* Willingness to participate in the entire study process, completing all examinations, surveys, and cost recordings as required.
* Ability to maintain contact throughout the study, with a fixed address and contact information.

Exclusion Criteria:

* Other eye conditions: history of strabismus, amblyopia, anisometropia, fundus diseases, dry eye, etc.
* Allergies: history of allergies to certain materials or medications.
* Surgical history: recent eye surgery.
* Non-compliance with required wear, follow-up, or lack of cooperation.
* Severe psychological disorders or behavioral problems.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population comprises children and adolescents aged 13-17 years with myopia ranging from -1.00D to -6.00D and astigmatism less than ±1.5D. Participants are first-time wearers of either peripheral defocus spectacles, single-vision frame glasses, or orthokeratology lenses. They are willing and able to complete all study requirements, including examinations, surveys, and cost recordings, and can maintain contact throughout the study duration with a stable address and contact information.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Quality of Life Scores | 1-Month Follow-up,3-Month Follow-up,6-Month Follow-up,12-Month Follow-up
  Improvement in Quality of Life Scores: The study will assess the impact of peripheral defocus spectacles, regular frame glasses, and orthokeratology lenses on the improvement of quality of life in myopic children and adolescents. This will be measured using the 'Pediatric Vision-Related Quality of Life Questionnaire' at baseline, 12 months post-treatment to evaluate and compare the long-term effects of these correction methods on quality of life."
Cost-Effectiveness Analysis | 1-Month Follow-up,3-Month Follow-up,6-Month Follow-up,12-Month Follow-up
  Cost-Effectiveness Analysis: This secondary outcome will assess the cost-effectiveness of peripheral defocus spectacles, regular frame glasses, and orthokeratology lenses in treating myopia in children and adolescents. The analysis will include the costs of acquiring, maintaining, and replacing these vision correction methods over a period of 12 months. This evaluation aims to provide a comprehensive financial comparison of these methods in terms of long-term expenditure and effectiveness in myopia management.

SECONDARY OUTCOMES:
Clinical Effectiveness Analysis | Baseline,1-Month Follow-up,3-Month Follow-up,6-Month Follow-up,12-Month Follow-up
  "Clinical Effectiveness Analysis: The study will evaluate the differences in vision correction effectiveness among peripheral defocus spectacles, regular frame glasses, and orthokeratology lenses in myopic children and adolescents. This includes vision tests (such as standard visual acuity charts) and ocular assessments to measure changes in axial length. These evaluations will be conducted at baseline, 6 months, and 12 months post-treatment to compare and analyze the clinical effectiveness of the various correction methods.

CONTACTS AND LOCATIONS:
Overall Officials: ruyi Li, Principal Investigator — He Eye Hospital
Locations (1):
- HeEyeHospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fricke TR, Jong M, Naidoo KS, Sankaridurg P, Naduvilath TJ, Ho SM, Wong TY, Resnikoff S. Global prevalence of visual impairment associated with myopic macular degeneration and temporal trends from 2000 through 2050: systematic review, meta-analysis and modelling. Br J Ophthalmol. 2018 Jul;102(7):855-862. doi: 10.1136/bjophthalmol-2017-311266. Epub 2018 Apr 26. PMID 29699985
- [Background] Ma Y, Qu X, Zhu X, Xu X, Zhu J, Sankaridurg P, Lin S, Lu L, Zhao R, Wang L, Shi H, Tan H, You X, Yuan H, Sun S, Wang M, He X, Zou H, Congdon N. Age-Specific Prevalence of Visual Impairment and Refractive Error in Children Aged 3-10 Years in Shanghai, China. Invest Ophthalmol Vis Sci. 2016 Nov 1;57(14):6188-6196. doi: 10.1167/iovs.16-20243. PMID 27842160
- [Background] Pan CW, Ramamurthy D, Saw SM. Worldwide prevalence and risk factors for myopia. Ophthalmic Physiol Opt. 2012 Jan;32(1):3-16. doi: 10.1111/j.1475-1313.2011.00884.x. PMID 22150586
- [Background] Pan CW, Wu RK, Li J, Zhong H. Low prevalence of myopia among school children in rural China. BMC Ophthalmol. 2018 Jun 11;18(1):140. doi: 10.1186/s12886-018-0808-0. PMID 29890943
- [Background] Dolgin E. The myopia boom. Nature. 2015 Mar 19;519(7543):276-8. doi: 10.1038/519276a. No abstract available. PMID 25788077
- [Background] Li Y, Liu J, Qi P. The increasing prevalence of myopia in junior high school students in the Haidian District of Beijing, China: a 10-year population-based survey. BMC Ophthalmol. 2017 Jun 12;17(1):88. doi: 10.1186/s12886-017-0483-6. PMID 28606071
- [Background] Wang J, Ying GS, Fu X, Zhang R, Meng J, Gu F, Li J. Prevalence of myopia and vision impairment in school students in Eastern China. BMC Ophthalmol. 2020 Jan 2;20(1):2. doi: 10.1186/s12886-019-1281-0. PMID 31898504
- [Background] Wu PC, Huang HM, Yu HJ, Fang PC, Chen CT. Epidemiology of Myopia. Asia Pac J Ophthalmol (Phila). 2016 Nov/Dec;5(6):386-393. doi: 10.1097/APO.0000000000000236. PMID 27898441
- [Background] Ma JX, Tian SW, Liu QP. Effectiveness of peripheral defocus spectacle lenses in myopia control: a Meta-analysis and systematic review. Int J Ophthalmol. 2022 Oct 18;15(10):1699-1706. doi: 10.18240/ijo.2022.10.20. eCollection 2022. PMID 36262865
- [Background] Yang T, Hu R, Tian W, Lin Y, Lu Y, Liang X, Zheng D, Zhang X. Comparison of Functional Vision and Eye-Related Quality of Life between Myopic Children Treated with Orthokeratology and Single-Vision Spectacles in Southern China. J Ophthalmol. 2023 Apr 8;2023:7437935. doi: 10.1155/2023/7437935. eCollection 2023. PMID 37089412
- [Background] Yang B, Ma X, Liu L, Cho P. Vision-related quality of life of Chinese children undergoing orthokeratology treatment compared to single vision spectacles. Cont Lens Anterior Eye. 2021 Aug;44(4):101350. doi: 10.1016/j.clae.2020.07.001. Epub 2020 Jul 13. PMID 32674999
- [Background] Walline JJ, Gaume A, Jones LA, Rah MJ, Manny RE, Berntsen DA, Chitkara M, Kim A, Quinn N. Benefits of contact lens wear for children and teens. Eye Contact Lens. 2007 Nov;33(6 Pt 1):317-21. doi: 10.1097/ICL.0b013e31804f80fb. PMID 17993828
- [Background] Walline JJ, Bailey MD, Zadnik K. Vision-specific quality of life and modes of refractive error correction. Optom Vis Sci. 2000 Dec;77(12):648-52. doi: 10.1097/00006324-200012000-00011. PMID 11147734